CLINICAL TRIAL: NCT04149808
Title: Comparative Prospective Study of Mepilex Ag vs. Xeroform in Pediatric Patients That Sustain Partial Thickness Burn Injury
Brief Title: Mepilex Ag vs. Xeroform in Pediatric Patients That Sustain Partial Thickness Burn Injury
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never conducted and no parcipants were ever enrolled and study never initiated.
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Elika Ridelman, Research Associate, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 061019MP2E
Record Dates: First submitted 2019-06-25; First posted 2019-11-04 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2019-10

CONDITIONS: Second-degree Burn

STUDY DESIGN:
Intervention Model Description: Patients under age 18 presenting to Children's Hospital of Michigan burn center or burn clinic with partial thickness, second degree scald burns.The burn must be at least 1% total body surface area (TBSA) or greater. The burn is divided approximately in half, with 50% of the wound receiving xeroform dressing and the remaining 50% receiving Mepilex Ag. Patients must present within 48 hours of injury. Patients must have a signed consent form (and oral assent for patients ages 7-12 or written assent for patients 13 years of age or greater).
Who Masked: Participant
Masking Description: The study was never initiated and study was terminated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Xeroform Control (Active Comparator): A single wound is treated with both the control (xeroform dressing) and intervention (Mepilex Ag). Approximately 50% of the wound is treated with xeroform dressing, which is the standard of care.
  Interventions: Device: Xeroform Dressing
- Mepilex Ag Intervention (Experimental): A single wound is treated with both the control (xeroform dressing) and intervention (Mepilex Ag). Approximately 50% of the wound is treated with Mepilex Ag; the product being tested.
  Interventions: Device: Mepilex Ag (burn dressing)

INTERVENTIONS:
Device: Mepilex Ag (burn dressing) — Dressing for low to medium exuding burns and wounds.
  Arms: Mepilex Ag Intervention
Device: Xeroform Dressing — Standard of care dressing for low to medium exuding burns and wounds.
  Arms: Xeroform Control

SUMMARY:
Pediatric patients that sustain partial thickness burn injuries to their extremities require regular scheduled dressings and weekly appointments for better healing. Typically, the dressing used at Children's Hospital of Michigan is Xeroform, which can often be painful when changing at the weekly clinic appointment. Mepilex Ag is also an approved treatment for these types of burns and has the potential to cause less pain with dressing changes, however is not used as frequently due to a much higher cost. Studies evaluating the treatment of partial thickness burns in pediatric patients have shown decreased cost and length of stay associated with dressings that are silver impregnated, like Mepilex Ag. However, these studies are all retrospective with a possible selection bias to patients. In addition, several studies have suggested less pain with newer foam and hydrofiber dressings. We are conducting a prospective study using patients with partial thickness burns of their extremities, applying Xeroform on half of the burn, and Mepilex Ag on the other half of the burn, to remove confounding variables between patients to determine the optimal burn dressing for partial thickness scald burns for pediatric patients. A partial thickness burn, also known as a second degree burn, extends into the top two layers of the skin, not passing the hypodermis. Our goal is to determine if Xeroform or Mepilex Ag is superior treatment for partial thickness burns in pediatric patients for healing time, appearance of scar, and patient pain and comfort during treatment and dressing changes.

DETAILED DESCRIPTION:
The patients will be recruited at the Children's Hospital of Michigan burn center or clinic by research personnel. If a patient is determined to fit inclusion criteria, parental consent will be obtained using the attached consent form by one of the research personnel. If the parent speaks another language, written consent will be obtained after explanation of the study and a short consent form in the native language. Also, a translator will be used to explain the full consent form used for English speaking patients. This form will be witnessed by a person who speaks the native language fluently. Only one parent will be required to sign consent as many patients only have one parent available in the hospital with them and this study involves only treatments that are current standard of care. If the patient is ages 7-12 years, an oral assent will be completed before participation in the study. If the patient is between ages 13-17, an assent form will be explained to them and their signature required to participate in the study. If they speak another language, assent will be obtained using a translator and the same methods listed above for parental consent. If the recruitment accrues beyond 4-6 non-english speaking participants, who speak a certain language, the consent forms will be translated into this language for future participants.

Study Protocol:

Once consent is obtained, and the patient is determined to be ready for a dressing application, one half of the extremity burn will be treated with Mepilex Ag and the other half of the extremity burn will be treated with Xeroform. Both of these treatments are current standard of care for a partial thickness scald burn in pediatric patients. The patients will be followed inpatient until they are discharged and then followed weekly at burn clinic appointments, the same care all of our burn patients receive. A survey will be administered to burn staff and patient's parents when the treatments are applied, at follow-up clinic appointments, and after the wound is healed completely. We will evaluate clinician and nurse ease of use, comfort of each dressing for the child, pain and itching associated with each dressing and dressing change, healing time, appearance of the scar after it is completely healed using the Vancouver Scar Scale, and parental satisfaction and ease of use for each dressing.

Data Collection and Evaluation:

A chart review will be performed for all patients to obtain demographic data including age, name, birth date, date of injury, injury details, the initial treatment applied if a different dressing was used before the patient was ready for application of Xeroform or Mepilex Ag, and any other pertinent information regarding the burn treatment. Study personnel and an attending physician will evaluate each patient at weekly follow-up visits or inpatient if the patient is being treated in the hospital. Survey results and other data will be evaluated after 10 patients complete treatment. Photographs taken as part of every burn patient's care may be reviewed as part of the study. These are obtained by medical photography and securely stored digitally. The Vancouver Scar Scale will be used for final evaluation of the healed scar after treatment is complete.

All data obtained in paper form will be stored in a locked filing cabinet in a locked office in the Pediatric Surgery Department and data obtained in digital form will be secure in a password protected file on the electronic medical record server.

Statistics will be performed using Statistical Package for Social Sciences (IBM version 22.0) and the statistical program R (r-project.org). The statistics to be performed for continuous variables (which are most of the assessment measures) will include a dependent groups analysis (e.g. paired samples t-test or robust analogue of this test such as Yuen's method for trimmed means, comparing medians, or bootstrap methods). The statistics to be performed for dichotomous measures will be the Sign test, which assesses differences in positive and negative outcomes for each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Patients under age 17 presenting to Children's Hospital of Michigan burn center or burn clinic with partial thickness, second degree scald burns to extremities.
* Burn of 1% TBSA or greater
* Within 48 hours of injury.
* Signed consent form (and oral assent for patients ages 7-12 or written assent for patients 13 years of age or greater).

Exclusion Criteria:

* Flame burns
* age over 18 years
* infection
* skin graft or donor site
* burns greater than 48 hours old.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Scar Evaluation | burn injury healing time; up to 10 weeks
  Vancouver Scar Scale: 0 is defined as normal in all instances
  * Vascularity: 0 to 3
  * Pigmentation: 0 to 3
  * Pliability/Elasticity: 0 to 5
  * Height: 0 to 3
  * Pain: 0 to 2
  * Itchiness: 0 to 2

SECONDARY OUTCOMES:
Dressing Change Survey | during the burn injury treatment, up to 10 weeks
  * Ease of application: 1 to 3; 3 is easiest
  * Pain during application: 1 to 10; 10 is most painful

CONTACTS AND LOCATIONS:
Overall Officials: Elika Ridelman, PhD, Study Director — Wayne State University
Locations (1):
- Children's Hospital of Michigan, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bugmann P, Taylor S, Gyger D, Lironi A, Genin B, Vunda A, La Scala G, Birraux J, Le Coultre C. A silicone-coated nylon dressing reduces healing time in burned paediatric patients in comparison with standard sulfadiazine treatment: a prospective randomized trial. Burns. 1998 Nov;24(7):609-12. doi: 10.1016/s0305-4179(98)00095-3. PMID 9882058
- [Background] Dykes PJ, Heggie R. The link between the peel force of adhesive dressings and subjective discomfort in volunteer subjects. J Wound Care. 2003 Jul;12(7):260-2. doi: 10.12968/jowc.2003.12.7.26567. PMID 12894697
- [Background] Gotschall CS, Morrison MI, Eichelberger MR. Prospective, randomized study of the efficacy of Mepitel on children with partial-thickness scalds. J Burn Care Rehabil. 1998 Jul-Aug;19(4):279-83. doi: 10.1097/00004630-199807000-00002. PMID 9710723
- [Background] Hollinworth H, Collier M. Nurses' views about pain and trauma at dressing changes: results of a national survey. J Wound Care. 2000 Sep;9(8):369-73. doi: 10.12968/jowc.2000.9.8.26282. PMID 11933365
- [Background] O'Donovan DA, Mehdi SY, Eadie PA. The role of Mepitel silicone net dressings in the management of fingertip injuries in children. J Hand Surg Br. 1999 Dec;24(6):727-30. doi: 10.1054/jhsb.1999.0270. PMID 10672813
- [Background] Platt AJ, Phipps A, Judkins K. A comparative study of silicone net dressing and paraffin gauze dressing in skin-grafted sites. Burns. 1996 Nov;22(7):543-5. doi: 10.1016/0305-4179(96)00035-6. PMID 8909755
- [Background] Williams G, Withey S, Walker CC. Longstanding pigmentary changes in paediatric scalds dressed with a non-adherent siliconised dressing. Burns. 2001 Mar;27(2):200-2. doi: 10.1016/s0305-4179(00)00082-6. PMID 11226664
- [Background] Winter GD (1975) Methods for the biological evaluation of dressings. In: Turner TD, Brain KR, eds. Surgical Dressings in the Hospital Environment. Surgical Dressings Research Unit, UWIST, Cardiff: 47-81
- See also: Pain at wound dressing change — https://ewma.org/fileadmin/user_upload/EWMA.org/Position_documents_2002-2008/position_doc2002_ENGLISH.pdf
- See also: Tool for assessing pain during dressing changes — http://www.worldwidewounds.com/2005/august/Hollinworth/Framework-Assessing-Pain-Wound-Dressing-Related.html
- See also: Descriptions of non-adherent dressings, their classification, and benefits — http://www.worldwidewounds.com/2003/